CLINICAL TRIAL: NCT00823901
Title: A Double-Blind, Placebo-Controlled, Pilot Study to Determine the Safety and Efficacy of Clindamycin Phosphate 1.2% and Tretinoin 0.025% Gel For The Treatment of Rosacea Over 12 Weeks
Brief Title: Safety and Efficacy Study of Clindamycin Phosphate 1.2% and Tretinoin 0.025% Gel to Treat Rosacea
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Medicis Pharmaceutical Corporation (Industry)
Responsible Party: Principal Investigator, Alexandra Kimball, Director, Clinical Unit for Research Trials in Skin, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008-P-001828
Record Dates: First submitted 2009-01-14; First posted 2009-01-16 (Estimated); Results first posted 2012-06-15 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Rosacea
Keywords: rosacea; clindamycin; tretinoin; clinical study; treatment
MeSH Terms: conditions — Rosacea | interventions — clindamycin phosphate; Tretinoin; Gels; clindamycin, tretinoin drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clindamycin/Tretinoin Gel (Experimental): Participants applied Clindamycin Phosphate 1.2% And Tretinoin 0.025% Gel on entire face (forehead, nose, chin, cheeks) once daily at night for 12 weeks
  Interventions: Drug: Clindamycin Phosphate 1.2% And Tretinoin 0.025% Gel
- Placebo gel (Placebo Comparator): Participants applied Placebo gel with no active medication on entire face (forehead, nose, cheeks, chin) once daily at night for 12 weeks.
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: Clindamycin Phosphate 1.2% And Tretinoin 0.025% Gel — Applied on entire face (forehead, nose, cheeks, chin) once daily at night for 12 weeks
  Other Names: Ziana
  Arms: Clindamycin/Tretinoin Gel
Drug: Placebo gel — Applied placebo gel with no active medication to entire face (forehead, nose, cheeks, chin) once daily at night for 12 weeks
  Other Names: placebo
  Arms: Placebo gel

SUMMARY:
The purpose of this study is to determine whether Clindamycin Phosphate 1.2% And Tretinoin 0.025% Gel are effective and safe in the treatment of papulopustular rosacea.

DETAILED DESCRIPTION:
Currently, there is no known cure for rosacea. The most effective treatment is systemic antibiotics, particularly of the tetracycline family. Topical treatments include metronidazole, antibacterials such as erythromycin and clindamycin, sulfacetamide and benzoyl peroxide. Isotretinoin (Accutane) is also used.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18 years of age and older.
2. Clinical diagnosis of papulopustular facial rosacea.
3. A minimum of 4 but not more than 50 facial inflammatory lesions (papules plus pustules).
4. Willing and able to understand and sign informed consent.
5. Able to complete study and comply with study procedures.

Exclusion Criteria:

1. Acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne, etc.), or severe acne requiring systemic treatment.
2. History or presence of regional enteritis or inflammatory bowel disease (e.g., ulcerative colitis, pseudomembranous colitis, chronic diarrhea, or a history of antibiotic-associated colitis, bloody diarrhea) or similar symptoms.
3. Use of topical rosacea treatments in the past 2 weeks.
4. Use of systemic antibiotics in the past 4 weeks.
5. Use of systemic retinoids within the past 3 months.
6. Use of laser or light based rosacea treatments within the past 2 months.
7. Concomitant use of medications that are reported to exacerbate rosacea, such as topical and systemic steroids as these may impact assessments.
8. Current drug or alcohol abuse.
9. Other dermatologic conditions that require the use of interfering topical or systemic therapy or that might interfere with study assessments such as, but not limited to, atopic dermatitis, perioral dermatitis or acne vulgaris.
10. Clinically significant abnormal findings or conditions (other than rosacea), which might, in the opinion of the Investigator, interfere with study evaluations or pose a risk to subject safety during the study.
11. Subjects who are pregnant or planning a pregnancy.
12. Use of any investigational therapy within the past 4 weeks.
13. Known hypersensitivity or previous allergic reaction to clindamycin or retinoids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2009-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexa Kimball, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Department of Dermatology - Stanford School of Medicine, Stanford, California
  - CURTIS - Massachussetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Background] Pelle MT, Crawford GH, James WD. Rosacea: II. Therapy. J Am Acad Dermatol. 2004 Oct;51(4):499-512; quiz 513-4. doi: 10.1016/j.jaad.2004.03.033. PMID 15389184
- [Background] Wilkin J, Dahl M, Detmar M, Drake L, Liang MH, Odom R, Powell F; National Rosacea Society Expert Committee. Standard grading system for rosacea: report of the National Rosacea Society Expert Committee on the classification and staging of rosacea. J Am Acad Dermatol. 2004 Jun;50(6):907-12. doi: 10.1016/j.jaad.2004.01.048. No abstract available. PMID 15153893
- [Background] Wilkin J, Dahl M, Detmar M, Drake L, Feinstein A, Odom R, Powell F. Standard classification of rosacea: Report of the National Rosacea Society Expert Committee on the Classification and Staging of Rosacea. J Am Acad Dermatol. 2002 Apr;46(4):584-7. doi: 10.1067/mjd.2002.120625. No abstract available. PMID 11907512
- [Background] Wilkin JK, DeWitt S. Treatment of rosacea: topical clindamycin versus oral tetracycline. Int J Dermatol. 1993 Jan;32(1):65-7. doi: 10.1111/j.1365-4362.1993.tb00974.x. PMID 8425809
- [Background] Diaz BV, Lenoir MC, Ladoux A, Frelin C, Demarchez M, Michel S. Regulation of vascular endothelial growth factor expression in human keratinocytes by retinoids. J Biol Chem. 2000 Jan 7;275(1):642-50. doi: 10.1074/jbc.275.1.642. PMID 10617662
- [Derived] Chang AL, Alora-Palli M, Lima XT, Chang TC, Cheng C, Chung CM, Amir O, Kimball AB. A randomized, double-blind, placebo-controlled, pilot study to assess the efficacy and safety of clindamycin 1.2% and tretinoin 0.025% combination gel for the treatment of acne rosacea over 12 weeks. J Drugs Dermatol. 2012 Mar;11(3):333-9. PMID 22395584

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at MGH and Stanford University Hospital.
Pre-assignment Details: Some subjects required a wash-out of medications they were using. Subjects were excluded if they did not have enough lesions.
Groups:
- Clindamycin/Tretinoin Gel: Participants applied Clindamycin Phosphate 1.2% And Tretinoin 0.025% Gel on entire face (forehead, nose, cheeks, chin) once daily at night for 12 weeks
- Placebo Gel: Participants applied Placebo vehicle gel (with out active ingredient) on entire face (forehead, nose, cheek, chin) once daily at night for 12 weeks
Period: Overall Study
Arm/Group | Clindamycin/Tretinoin Gel | Placebo Gel
Started | 43 (Randomized to clindamycin/tretinoin gel) | 40 (Randomized to placebo gel)
Completed | 39 (Discontinued intervention (n=2) Only baseline completed (n=2)) | 38 (Discontinued intervention (n=1) Only baseline completed (n=1))
Not Completed | 4 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clindamycin/Tretinoin Gel | Placebo Gel | Total
Number analyzed (Participants) | 43 | 40 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 39 | 81
  >=65 years | 1 | 1 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 53.2 (13.6) | 51.2 (14.0) | 52.17 (13.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 31 | 59
  Male | 15 | 9 | 24
Region of Enrollment [Number; unit: participants]
  United States | 43 | 40 | 83

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Number of Inflammatory Lesions From Baseline to Week 12
Description: The number of inflammatory lesions (papules and pustules) on the face were counted by a dermatologist at baseline and week 12 for each participant. Change in the number of inflammatory lesions is defined as week 12 values minus the baseline values of the participant. Last observation carried forward (LOCF) method was used for missing values.
Time Frame: Baseline, week 12
Population: Intent to treat (ITT) population. Participants who were randomized but only had baseline visit (never began treatment) were excluded from the analysis. Last observation carried forward (LOCF) was also used.
Measure: Mean (Standard Deviation); unit: lesions
Groups:
- Placebo: Participants applied placebo gel without active ingredient on entire face (forehead, nose, cheek, chin)once daily at night for 12 weeks
Arm/Group | Clindamycin/Tretinoin Gel | Placebo
Number analyzed (Participants) | 41 | 39
lesions | .83 (10.84) | -3.13 (13.28)
Statistical Analysis 1: Comparison: Clindamycin/Tretinoin Gel vs Placebo; Test type: Superiority or Other; p = 0.15, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 weeks (duration of study participation)
Arm/Group | Clindamycin/Tretinoin Gel | Placebo Gel
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/40
Other Adverse Events (participants affected / at risk) | 29/41 | 11/39
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clindamycin/Tretinoin Gel (N=41) | Placebo Gel (N=39)
Worsening rosacea (Skin and subcutaneous tissue disorders) | 7 (7) | 4 (4)
Facial scaling (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)
Facial Dryness (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)
Facial redness (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Facial burning sensation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Facial itching (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Facial irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
This study is limited by relatively small number of subjects. In addition, overall assessment of acne rosacea severity as determined by subjects' self-assessment was not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No